CLINICAL TRIAL: NCT06030349
Title: Real World Clinical Outcomes From Treatment and Evaluation of Obstructive Sleep Apnoea Syndrome in Children With Down Syndrome
Brief Title: Clinical Outcomes From Treatment and Evaluation of Obstructive Sleep Apnoea in Children With Down Syndrome
Acronym: REFRESHED
Status: Recruiting | Type: Observational
Sponsor: Children's Health Ireland (Other Government)
Collaborators: University of Edinburgh (Other); Birmingham Children's Hospital (Other); Belfast Health and Social Care Trust (Other); University Hospital Southampton NHS Foundation Trust (Other); University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Sheila Javadpour, Clinical Lead for Respiratory Sleep Medicine, Children's Health Ireland
Other Study IDs: REC137-22
Record Dates: First submitted 2023-04-30; First posted 2023-09-11 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Obstructive Sleep Apnea; Down Syndrome; Quality of Life; Behavior; Adherence, Treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive; Down Syndrome; Behavior; Treatment Adherence and Compliance | interventions — Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Standard: In addition to data from clinical assessment, sleep studies and non-invasive ventilator downloads recorded as part of standard care participants will undergo questionnaire assessment of behaviour, quality of life and barriers to tolerating treatment. Participants aged 3 years and above will receive the Child Sleep Habits Questionnaire, Obstructive Sleep Apnoea-18 questionnaire and Adherence Barriers to CPAP (Continuous Positive Airway Pressure) Questionnaire. Participants aged 6 months to 3 years will receive the Brief Infant Sleep Questionnaire, Infant Toddler Quality of Life - Short Form 47, Obstructive Sleep Apnoea -18 Caregiver Concern Domain and a modified version of the Adherence Barriers to CPAP Questionnaire.
  Interventions: Device: Non-invasive ventilation
- Advanced: In addition to all elements of the standard testing group, a sub-group of up to 20 participants will be invited to take part in 45-60 minute semi-structured interviews exploring expectations, experiences and barriers encountered.
  Interventions: Device: Non-invasive ventilation

INTERVENTIONS:
Device: Non-invasive ventilation — Non-invasive ventilation

SUMMARY:
The goal of this observational study is to learn about the use of non-invasive ventilation for treatment of obstructive sleep apnoea syndrome in children with Down Syndrome. The main questions it aims to answer are:

* What is the impact of non-invasive ventilation on sleep behaviours and quality of life?
* What barriers are faced by children and their families in establishing tolerance to non-invasive ventilation?

Participants will be asked to complete questionnaires before and after starting treatment. Researchers will compare this data with the results of sleep studies and non-invasive ventilator downloads recorded as part of standard medical care. A sub-group of up to 20 participants will be invited to take part in 45-60 minute interviews exploring expectations, experiences and barriers encountered during non-invasive ventilation therapy.

DETAILED DESCRIPTION:
Our aim is to examine the impact of non-invasive ventilation for treatment of obstructive sleep apnoea syndrome in children with Down Syndrome on behavioural and quality of life outcomes and to establish the specific barriers experienced in establishing adherence to treatment.

Information from clinical assessment, sleep studies and device downloads recorded as part of standard care will be combined with questionnaire data to assess for changes in behaviour and quality of life. All participants will undergo questionnaire assessment of barriers experienced. A sub-group of up to 20 participants will be invited to take part in 45-60 minute semi-structured interviews exploring expectations, experiences and barriers encountered.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a confirmed diagnosis of Down Syndrome where a clinical decision has been made to initiate respiratory support with non-invasive ventilation.
* Obstructive Apnoea Hypopnoea Index > 2 episodes/hour or where sleep disordered breathing symptoms occur in combination with an Apnoea Hypopnoea Index > 1 episode/hr. - English language proficiency.
* Age ≥ 4 months at the commencement of therapy.

Exclusion Criteria:

* Individuals not willing to comply with study procedures or assessments.
* Individuals for whom ventilatory support devices are already prescribed and those with artificial airways.
* Individuals on clinical trials of investigational support therapies.

Ages: 6 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with Down Syndrome referred for evaluation for suspected sleep disordered breathing
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-11-28 (Actual); Primary Completion 2027-11-28 (Estimated); Study Completion 2027-12-28 (Estimated)

PRIMARY OUTCOMES:
To determine the effect of treatment of obstructive sleep apnoea syndrome with non-invasive ventilation on quality of life in children with Down Syndrome > 3 years. | Prior to and following 8 weeks attempted initiation of non-invasive ventilation treatment
  Change in Obstructive Sleep Apnoea - 18 scores (Range 0- 126, Higher scores indicating worse quality of life) from baseline will be used to evaluate for improvement in sleep related breathing specific quality of life in children >3 years. Sleep disturbance, physical suffering, emotional distress, daytime problems and caregiver concern subscales will also be evaluated for change.
To determine the effect of treatment of obstructive sleep apnoea syndrome with non-invasive ventilation on quality of life in children with Down Syndrome < 3 years. | Prior to and following 8 weeks attempted initiation of non-invasive ventilation treatment
  Change in Infant Toddler Quality of Life - Short Form 47 scores (Range 0 - 100, Higher scores indicating greater quality of life) from baseline will be used to evaluate for improvement in sleep related breathing specific quality of life in children < 3 years. Infant and parent subscales will also be evaluated for change.
To determine the effect of treatment of obstructive sleep apnoea syndrome with non-invasive ventilation on caregiver concerns regarding sleep disordered breathing for caregivers of children with Down Syndrome < 3 years. | Prior to and following 8 weeks attempted initiation of non-invasive ventilation treatment
  Change in Caregiver-concern domain of the Obstructive Sleep Apnoea - 18 (Range 0 - 28, Higher scores indicating worse quality of life) from baseline will be used to evaluate for change in caregiver concern regarding sleep disordered breathing.
To determine the effect of treatment of obstructive sleep apnoea with non-invasive ventilation on sleep behaviours in children with Down Syndrome > 3 years. | Prior to and following 8 weeks attempted initiation of non-invasive ventilation treatment
  Change in Child Sleep Habits Questionnaire scores (Range 0 - 97, Higher scores indicating greater sleeping difficulties) from baseline will be used to evaluate for overall improvement in sleep behaviours in children > 3 years. Bedtime resistance, sleep onset delay, sleep duration, sleep anxiety, night waking, parasomnia, sleep disordered breathing and daytime sleepiness subscales will also be evaluated for change.
To determine the effect of treatment of obstructive sleep apnoea with non-invasive ventilation on sleep behaviours in children with Down Syndrome < 3 years. | Prior to and following 8 weeks attempted initiation of non-invasive ventilation treatment
  Change in Brief Infant Sleep Questionnaire scores (Range 0 - 100, Lower scores indicating greater sleeping difficulties) from baseline will be used to evaluate for overall improvement in sleep behaviours in children < 3 years. Infant sleep, parent perception and parent behaviour subscales will also be evaluated for change.
To establish the specific barriers to adherence faced by children > 3 years with Down Syndrome and their caregivers when starting non-invasive ventilation for the treatment of obstructive sleep apnoea syndrome | Prior to and following 8 weeks attempted initiation of non-invasive ventilation treatment
  Quantitative assessment of barriers encountered in establishing adherence will be evaluated using the Continuous Positive Airway Pressure Questionnaire (Range 29-145, Higher scores indicating greater barriers to adherence) for children > 3 years. Behaviours/belief/environment, emotional and physical subscales will also be evaluated for change.
To establish the specific barriers to adherence faced by children < 3 years with Down Syndrome and their caregivers when starting non-invasive ventilation for the treatment of obstructive sleep apnoea syndrome | Prior to and following 8 weeks attempted initiation of non-invasive ventilation treatment
  Quantitative assessment of barriers encountered in establishing adherence will be evaluated using the Modified Continuous Positive Airway Pressure Questionnaire (Range 27 - 135, Higher scores indicating greater barriers to adherence) for children < 3 years. This is a non-validated questionnaire developed by our research group.
Assessment of expectations, experiences and barriers experienced by families in the treatment of obstructive sleep apnoea syndrome with non-invasive ventilation | After 8 weeks of attempted initiation of non-invasive ventilation
  Qualitative assessment of expectations, experiences and barriers experienced during non-invasive ventilation treatment will be explored through semi-structured interviews to add nuance to the outcomes around efficacy of treatment, quality of life, behaviour, and treatment adherence

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Javadpour, Principal Investigator — Children's Health Ireland
Locations (6):
- Ireland (2):
  - Trinity College Dublin, Dublin
  - Children's Health Ireland, Dublin
- United Kingdom (4):
  - Royal Belfast Hospital for Sick Children, Belfast
  - Birmingham Children's Hospital, Birmingham
  - Royal Hospital for Children & Young People, Edinburgh
  - Southampton Children's Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No